CLINICAL TRIAL: NCT06304610
Title: Hospital-based Validation of the New ELEVATE Screening Tool in Belgium and Ecuador
Brief Title: Hospital-based Validation of the New ELEVATE Screening Tool
Acronym: ELEVATE-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Horizon 2020 - European Commission (Other); Universidad de Cuenca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0044
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer; HPV Infection
Keywords: cervical cancer; screening; self-sampling; HPV; underscreened; new ELEVATE tool
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: all participants receive the same tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sample taking and questionnaire (Experimental): The participant is invited in the colposcopy waiting room by the study nurse and is asked to follow the study nurse to a separate room. Here the participant is given all the information about the study and sampling. If the participant agrees to participate and signs the consent form, the study nurse registers the participant and then asks her to complete a very short questionnaire. After that, the participant will be asked to take a self-sample.
  Then the participant will proceed to her appointment for colposcopy. The doctor will take an endocervical samples, similar to a pap smear, before the actual colposcopy examination begins. Her samples will then be analyzed with the newly developed ELEVATE test and with comparative lab tests (standard HPV DNA detection and protein detection tests) in order to validate the newly developed ELEVATE cervical cancer screening test.
  Participation is free and the participant can stop your participation at any time.
  Interventions: Behavioral: Questionnaire; Procedure: HPV self-sample; Procedure: Endocervical sample

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire to probe socio-demographic data and information regarding sexual and reproductive health.
Procedure: HPV self-sample — Collection of HPV self-sample. The study nurse will explain step by step how the participant should take the test. The participant will also be given written instructions and the study nurse will always be around if the participant has any questions. The participant will be asked to take the self-sample in a private room with toilet. After collection the sample is handed back to the study nurse, who will then take the samples to the laboratory for analysis.
Procedure: Endocervical sample — Endocervical sample taken by the gynaecologist. This procedure can be somewhat uncomfortable but not painful. The participant may always ask questions if she has any doubts or questions. The gynaecologist will perform the standard colposcopy examination after collection (for which the woman sits in the colposcopy waiting room)

SUMMARY:
ELEVATE is a six-year project, conducted by an international research alliance led by Ghent University, aiming to develop a new test and approach for cervical cancer screening in hard-to-reach populations.

In this final stage of the project, a hospital-based validation study is deployed in Belgium and Ecuador to clinically validate the new ELEVATE screening test based on self-samples and endocervical samples. The simultaneous detection of HPV DNA and the proteomic markers allows for the detection of those cervical HPV infections associated with progression towards cervical cancer.

At each study site, 100 women between 30-65 years old, with a recent abnormal pap smear result will be recruited in the colposcopy waiting room. After registration and signing the informed consent form, each woman will be asked to fill out a short self-administered questionnaire for socio-demographic information. Each woman will provide a self-sample as well as an endocervical sample before the colposcopy examination. Both samples of all 200 women (i.e. participants from Belgium and Ecuador) will be tested with the new ELEVATE screening test, using 400 ELEVATE cartridges, as well as with standard tests.

Besides analyzing all samples on the new ELEVATE screening test, the following standard tests will also be performed on all samples (at Ghent University - including the shipped samples of Ecuador):

* AnyplexTM II HPV HR Detection (Segeene Inc., Korea): approved comparison test
* ELISA protein detection: only available comparison test

In order to generate HPV DNA results locally, that can be communicated to the participants in short time (versus waiting for AnyplexTM II HPV HR Detection test results after shipment to Belgium), in Ecuador the following additional standard test will be performed on the100 endocervical samples (before shipment to Belgium):

• HPV DNA Mole Bioscience test

Concordance between the test results of the ELEVATE screening test and standard lab tests on both type of samples will be defined, for HPV DNA as well as protein detection. Additionally, the sensitivity and specificity of the HPV DNA test and the protein test of the ELEVATE screening test will be defined, according to clinically relevant outcomes.

DETAILED DESCRIPTION:
ELEVATE is a six-year project, conducted by an international research alliance led by Ghent University, aiming to develop a new test and approach for cervical cancer screening in hard-to-reach populations.

In this final stage of the project, a hospital-based validation study is deployed in Belgium and Ecuador to clinically validate the new ELEVATE screening test based on self-samples and endocervical samples. This point-of-care test is a portable, battery-powered device compatible with self-sampling and comprises a Human Papillomavirus (HPV) DNA test as well as a proteomic biomarkers detection sensor, aiming for high sensitivity and specificity. The test can be offered in a broad range of settings and results are available in less than 24 hours, eliminating the need for sample storage and lab infrastructure. The simultaneous detection of HPV DNA and the proteomic markers allows for the detection of those cervical HPV infections associated with progression towards cervical cancer.

At each study site, 100 women between 30-65 years old, with a recent abnormal pap smear result will be recruited in the colposcopy waiting room. After registration and signing the informed consent form, each woman will be asked to fill out a short self-administered questionnaire for socio-demographic information. Each woman will provide a self-sample as well as an endocervical sample before the colposcopy examination. The self-sample will be taken by using the Evalyn brush (Rovers - CE-approved device), while the endocervical sample will be taken by the gynaecologist with a standard endocervical brush used in the hospital. Both sampling measures are considered non-invasive. The ELEVATE screening tool is composed out of a device and cartridges. The ELEVATE cartridge is a microfluidic cartridge, consisting of the 2 sensor types (genomic and proteomic), onto which cervical fluid will be brought drop by drop. This cartridge will then be introduced into the ELEVATE screening device, after which via electrochemical signals the HPV DNA and protein result will become clear. The new ELEVATE screening test (or tool) is an HPV DNA detection and protein detection test under development; results based on the new test will not be shared with the patient or health care provider. Results of the tool will be compared with standard laboratory tests. Only the result of the standard laboratory tests will be fed back to the patient if requested by the patient (as also mentioned in the ICF).

The following tests will be performed at UZ Gent:

* new ELEVATE screening test (HPV DNA detection and protein detection) on self-sample and endocervical samples from women from Belgium (100 women, 200 samples)
* Standard lab test HPV DNA Detection: AnyplexTM II HPV HR Detection (Segeene Inc., Korea): approved comparison test; on all samples, including samples sent to Belgium from the women from Ecuador (200 women, 400 samples)
* Standard lab test protein detection: ELISA protein detection: only available comparison test; on all samples, inlcuding samples sent to Belgium from the women from Ecuador (200 women, 400 samples)

In order to generate HPV DNA results locally, that can be communicated to the participants in short time (versus waiting for AnyplexTM II HPV HR Detection test results after shipment to Belgium), in Ecuador the following additional standard test will be performed on the100 endocervical samples (before shipment to Belgium):

* HPV DNA Mole Bioscience test
* new ELEVATE screening test (HPV DNA detection and protein detection) on self-test and endocervical sample from women from Ecuador (100 women, 200 samples)

Concordance between the test results of the ELEVATE screening test and standard lab tests on both type of samples will be defined, for HPV DNA as well as protein detection. Additionally, the sensitivity and specificity of the HPV DNA test and the protein test of the ELEVATE screening test will be defined, according to clinically relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* have a previous abnormal pap smear/recent diagnosis of cervical dysplasia (<4 months) and therefore have a colposcopy appointment, or
* a positive HPV test (<4 months) and therefore have a colposcopy appointment, and
* able to understand the study materials (questionnaire) and informed consent form

Exclusion Criteria:

* women with heavy bleeding at consultation
* women with known pregnancy at consultation
* women who are undergoing or have completed chemotherapy in the six months prior to the enrollment, or received LEEP, cryotherapy or another treatment in the six months prior to enrollment
* women who do not consent

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical validation | Up to 8 months
  To determine the sensitivity and specificity of the new ELEVATE screening test, combining HPV DNA detection and biomarker detection, according to clinically relevant outcomes (coloscopy results).

SECONDARY OUTCOMES:
Concordance | Up to 8 months
  To determine the concordance between the test results of the new ELEVATE screening test and standard tests on the self-sample and endocervical sample (for both HPV DNA and protein detection).
HPV DNA test validation | Up to 8 months
  To determine the sensitivity and specificity of the HPV DNA test of the ELEVATE screening test according to clinically relevant outcomes
Protein test validation | Up to 8 months
  To determine the sensitivity and specificity of the protein test of the ELEVATE screening test according to clinically relevant outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Degomme, MD,PhD,Prof, Study Chair — International Centre of Reproductive Health; Philippe Tummers, MD,PhD,Prof, Principal Investigator — Vrouwenkliniek, UZ Ghent; Bernardo José Vega Crespo, MD, Principal Investigator — Universidad de Cuenca
Locations (2):
- Ghent University Hospital, Ghent, East-Flanders, Belgium
- SOLCA University Hospital, Cuenca, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: Related Info — https://elevate-hpv.com/